CLINICAL TRIAL: NCT06739200
Title: Evaluation of PRF Membrane in Postoperative Recovery: A Preliminary Study Using 3D Imaging in Periapical Surgery
Brief Title: PRF Membrane and Recovery After Periapical Surgery: A 3D Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3736-1/2022/EKU
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Periapical Diseases; Radicular Cyst; Granuloma; Postoperative Complications; Pain, Postoperative
MeSH Terms: conditions — Periapical Diseases; Radicular Cyst; Granuloma; Postoperative Complications; Pain, Postoperative | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Membrane Group (Experimental): Participants in this group will undergo periapical surgery in which a platelet-rich fibrin (PRF) membrane will be placed at the surgical site. The PRF membrane is designed to promote healing and reduce postoperative swelling and pain. Outcomes, including swelling, pain levels, and healing progress, will be evaluated.
  Interventions: Procedure: Platelet-Rich Fibrin (PRF) Membrane
- Control Group (No Intervention): Participants in this group will undergo periapical surgery without the use of a PRF membrane. This group will serve as a comparison to evaluate the effectiveness of the PRF membrane in promoting healing and reducing postoperative swelling and pain. Outcomes, including swelling, pain levels, and healing progress, will be evaluated.

INTERVENTIONS:
Procedure: Platelet-Rich Fibrin (PRF) Membrane — The Platelet-Rich Fibrin (PRF) membrane is a biocompatible material derived from the participant's own blood and prepared through centrifugation. It is applied at the surgical site during periapical surgery to promote tissue regeneration, enhance wound healing, and reduce postoperative swelling and pain. Unlike synthetic materials, PRF is autologous and does not require additional chemical additives or processing. This study aims to evaluate its effectiveness in improving recovery outcomes compared to surgery without PRF membrane placement.
  Arms: PRF Membrane Group

SUMMARY:
The goal of this clinical trial is to determine whether a PRF (platelet-rich fibrin) membrane helps improve recovery after periapical surgery in adults. The main questions it seeks to answer are:

Does the use of a PRF membrane reduce swelling and pain after surgery? Does the use of a PRF membrane improve healing as observed on 3D imaging? Researchers will compare the outcomes of participants who receive a PRF membrane during surgery with those who do not, to assess whether the PRF membrane improves recovery.

Participants will:

Undergo periapical surgery with or without the use of a PRF membrane. Have swelling and pain assessed at specific time points after surgery. Participate in 3D imaging scans to evaluate healing.

Participants will:

Undergo periapical surgery with or without the use of a PRF membrane. Have swelling and pain measured at specific time points after surgery. Take part in 3D imaging scans to evaluate healing.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-65 years, both male and female.
* Diagnosed with periapical disease, including periapical cysts or granulomas.
* Requiring periapical surgery as part of their treatment plan.
* Presenting a tooth needing endodontic surgery with periradicular lesions of strictly endodontic origin.
* Size of the bone crypt between 6 mm and 12 mm.
* Non-surgical retreatment considered unfeasible or previously failed.
* Apical root canal free from posts over a length of at least 6 mm.
* Adequate coronal restoration without coronal leakage.
* Willing and able to provide written informed consent.
* Capable of attending follow-up visits and participating in required assessments.
* Maxillary and mandibular teeth limited to the 2nd premolar to 2nd premolar regions.
* Without general medical contraindications for oral surgical procedures.

Exclusion Criteria:

* Patients with systemic conditions affecting healing, such as:

  * • Uncontrolled diabetes mellitus.
  * • Autoimmune disorders.
  * • Chronic inflammatory diseases.
* Pregnant or breastfeeding individuals.
* Use of medications or therapies that may interfere with healing, including:

  * • Bisphosphonates.
  * • Immunosuppressants.
  * • Radiotherapy.
  * • Oncological therapies (e.g., chemotherapy, immunotherapy).
* Requires antibiotic prophylaxis or therapy.
* History of allergies or adverse reactions to blood-derived products.
* Neuropsychiatric disorders.
* Active infection or severe periodontal disease in the surgical area.
* Periodontal probing depths greater than 5 mm.
* Moderate to severe periodontal bone loss.
* Vertical root fractures.
* Perforation of the furcation area or root canal, except for the apical area.
* Smokers or individuals unwilling to refrain from smoking during the study period.
* Participation in another clinical trial within the last 30 days.
* Absolute or relative contraindications for surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (QoL) Using the PROMIS-29+2 Profile v2.1 | Preoperative and Day 7 postoperative.
  Quality of life (QoL) was evaluated using the Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 questionnaire, a validated tool assessing health-related QoL across multiple domains, including physical function, emotional stress, sleep disturbance, and social tasks. Each domain is scored using a standardized T-score scale, ranging from 20 (lowest) to 80 (highest), where higher scores indicate better quality of life.
  Time Points: Preoperative and Day 7 postoperative.
  Unit of Measure: PROMIS T-score (range: 20-80).
Change in Pain Intensity Using the Visual Analog Scale (VAS) | Daily assessments from Day 0 (day of surgery) to Day 7 postoperative.
  Pain intensity was measured daily using the Visual Analog Scale (VAS), a validated tool for assessing patient-reported pain. The VAS scale ranges from 0 (no pain) to 10 (worst possible pain), where higher scores indicate worse pain outcomes. Measurements were taken daily for seven days following surgery.
  Time Points: Daily from Day 0 (day of surgery) to Day 7 postoperative.
  Unit of Measure: Scale Points (range: 0-10).
Change in Postoperative Swelling Using 3D Optical Scans | Measurements were taken at T0 (preoperative) and T1 (Day 3 postoperative).
  Postoperative swelling was measured volumetrically using 3D optical scans performed with the Einstar 3D scanner (Shining 3D, Hangzhou, China). Measurements were taken preoperatively (T0) and on Day 3 postoperative (T1). Swelling volume is expressed in cubic centimeters (cm³), where a higher volume indicates greater swelling.
  Time Points: Preoperative (T0) and Day 3 postoperative (T1).
  Unit of Measure: Cubic centimeters (cm³).

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Oral and Maxillofacial Surgery, Budapest, Mária Utca 52, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Major M, Meszaros B, Wursching T, Polyak M, Kammerhofer G, Nemeth Z, Szabo G, Nagy K. Evaluation of a Structured Light Scanner for 3D Facial Imaging: A Comparative Study with Direct Anthropometry. Sensors (Basel). 2024 Aug 15;24(16):5286. doi: 10.3390/s24165286. PMID 39204985

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT06739200/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT06739200/ICF_001.pdf